CLINICAL TRIAL: NCT05670860
Title: Comitial Prophylaxis in Neurosurgery in Patients Who Have Undergone Intracranial Surgery Programmed Supratentorial Surgery (Exeresis or Biopsy) Between 2019 and 2022
Acronym: PRO-CON
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC22.0198
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Anti-epileptic Prophylaxis in Intracranial Neurosurgery
Keywords: anti-epileptic prophylaxis; intracranial neurosurgery; epileptic seizures
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anti-epileptic prophylaxis: The first group consists of patients treated between January 2019 and late 2020 who were given systematic prophylaxis
- NO Anti-epileptic prophylaxis: Patients from the second group were treated between 2021 and 2022 and did not receive any prophylaxis

SUMMARY:
JUSTIFICATION Anti-epileptic prophylaxis has long been a systematic practice for supra-tentorial intracranial surgeries. Since 2021, European guidelines no longer recommend this prophylaxis and practices have evolved.

We therefore propose to compare epileptic seizure's occurrence in the first postoperative month between two groups of neurosurgical patients.The first group consists of patients treated between January 2019 and late 2020 who were given systematic prophylaxis. Patients from the second group were treated between 2021 and 2022 and did not receive any prophylaxis.

The secondary objective will consist in identifying the number of patients placed on prophylaxis, the length of prophylaxis, treatment's side effects (depression, elevated liver enzymes…), and comparing patients' neurological outcome at 3 and 6 months after surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years old
* Expressed non-opposition
* Patient who underwent supratentorial intracranial surgery (either resection or biopsy) at Brest University Hospital from January 01, 2019 to September 01, 2022.

Exclusion Criteria:

* Refusal to participate
* Patient under legal protection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients underwent a supratentorial intracerebral elective surgery (resection or biopsy) over the period from January 01, 2019 to September 01, 2022.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-05-22 (Estimated); Study Completion 2023-05-22 (Estimated)

PRIMARY OUTCOMES:
The number of epileptic seizures during the first postoperative month (between D-0 and D-30) of neurosurgery patients treated for elective supratentorial intracranial procedures. | the first postoperative month (between D-0 and D-30)

SECONDARY OUTCOMES:
Commencement of anti-epileptic treatment Length of prophylaxis Treatment's side effects Neurological outcome at 3 and 6 months (RANKIN modified score) | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.